CLINICAL TRIAL: NCT05282810
Title: Cartilage Versus Temporalis Fascia Graft in Tympanoplasty for Recurrent Tympanic Membrane
Brief Title: Cartilage Versus Temporalis Fascia Graft in Tympanoplasty for Recurrent Tympanic Membrane Perforation '' Comparative Study ''
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Caroleen Mounir Tawfik, researcher, Assiut University
Other Study IDs: recurrent tympanoplasty
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Tympanoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- cartilage tympanoplasty: use cartilage in tympanoplasty for recuurent perforation
  Interventions: Other: tympanoplasty
- temporalis fascia graft in tympanoplasty: use temporalis fascia as a graft in tympanoplasty for recuurent perforation
  Interventions: Other: tympanoplasty

INTERVENTIONS:
Other: tympanoplasty — use of cartilage versus tempotalis fascia in tympanoplasty for recuurent perforation

SUMMARY:
Use of Cartilage Versus Temporalis Fascia as a Graft in Tympanoplasty for Recurrent Tympanic Membrane Perforation

DETAILED DESCRIPTION:
The main aim of successful tympanoplasty is to create a well aerated closed cavity after total removal of the disease. Numerous types of grafting materials have been used for closure of the tympanic membrane including fascia, periosteum, perichondrium, cartilage, vein, skin, and fat tissue . Autografts are thought to be the most compatible grafting materials with the best surgical results in tympanoplasty Temporal muscle fascia is composed of irregularly arranged elastic fibers and fibrous connective tissue. For this reason postoperative dimensions of temporal muscle fascia are unpredictable.

Cartilage has a constant shape, firmer than fascia and also lack fibrous tissue, so that postoperative dimensions remains the same and beside this, it is also nourished by diffusion and show great adaptation with TM . These advantages make the cartilage graft more preferable by otologists recently.

the use of cartilage graft in many different ways such as perichondrium cartilage island technique, palisade technique or cartilage reinforcement technique

ELIGIBILITY:
Inclusion Criteria:

* patients with safe chronic suppurative otitis media patient with recurrent perforation patirnt with coductive hearing loss

Exclusion Criteria:

* sensorineural hearing loss active infection compromised immune system

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be randomly divided into Group 1, where only temporalis fascia alone will be used as a graft and Group 2, where cartilage will be used along with temporalis fascia graft.
  Patients will be followed up and examined at 2 and 6 month to assess
  1. graft take up (healing)
  2. pure tone audiometry( hearing )
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Cartilage Versus Temporalis Fascia Graft in Tympanoplasty for Recurrent Tympanic Membrane Perforation '' Comparative Study '' | Baseline
  compare of improvment of hearing by using temporalis fascia versus cartilage tympanoplasty in recurrent perforation compare of graft take up by using temporalis fascia versus cartilage tympanoplasty in recurrent perforation

REFERENCES:
- [Background] Jalali MM, Motasaddi M, Kouhi A, Dabiri S, Soleimani R. Comparison of cartilage with temporalis fascia tympanoplasty: A meta-analysis of comparative studies. Laryngoscope. 2017 Sep;127(9):2139-2148. doi: 10.1002/lary.26451. Epub 2016 Dec 9. PMID 27933630
- [Background] Shakya D, Nepal A. Long-term results of type I tympanoplasty with perichondrium reinforced cartilage palisade vs temporalis fascia for large perforations: A retrospective study. J Otol. 2021 Jan;16(1):12-17. doi: 10.1016/j.joto.2020.07.004. Epub 2020 Jul 29. PMID 33505444